CLINICAL TRIAL: NCT07032168
Title: Influence of Lifestyle Factors, Cardiorespiratory Fitness, and Body Composition on Plasma BDNF and pTau217 Levels and Cognitive Function in Healthy Young Adults
Brief Title: Lifestyle, Fitness, and Plasma Biomarkers in Healthy Young Adults
Acronym: NEUROACTIVE
Status: Recruiting | Type: Observational
Sponsor: European University Miguel de Cervantes (Other)
Responsible Party: Sponsor
Other Study IDs: PI-DOC010-NEUROACTIVE
Record Dates: First submitted 2025-05-26; First posted 2025-06-22 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy Young Adults
Keywords: Neuroplasticity; Lifestyle; Healthy young adults; Plasma biomarkers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy young adults: Healthy young adults (18-24 years old)

SUMMARY:
Lifestyle play a key role in modulating brain health by directly influencing a number of key biological processes, such as neuroplasticity, neurogenesis, and regulation of biomarkers associated with cognitive decline. Factors such as physical activity, diet, sleep quality, stress management, and body composition have been shown to have a significant impact on neuroprotection and cognitive performance. These factors not only contribute to maintaining metabolic and functional balance in the body, but are also linked to the expression of biomarkers such as brain-derived neurotrophic factor (BDNF) and Tau protein phosphorylated at the amino acid threonine 217 (PTau217), which are essential for the maintenance of neuronal health and the prevention of neurodegenerative diseases. In this sense, a healthy lifestyle, characterized by regular physical activity, a balanced diet, good quality sleep, low stress levels and adequate body composition, can act as a protective factor against cognitive decline from early stages of life.

ELIGIBILITY:
The following inclusion criteria are established:

1. Age between 18 and 24 years.
2. Not have chronic or neurodegenerative diseases.
3. Not be on pharmacological treatment that affects the central nervous system or metabolism.

The exclusion criteria for participants:

1. Medical or traumatological condition that makes it impossible to practice physical exercise.
2. Musculoskeletal injury within 6 months prior to the first visit to the laboratory.
3. Recent surgery (<3 months).
4. Have a medical condition in which physical activity is contraindicated (assessed with the Physical Activity Predisposition Questionnaire (PARQ+).

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults, between 18 and 24 years old.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Plasma biomarkers | Baseline
  Plasma concentrations of BDNF and pTau217 will be assessed using ELISA kits. Fasting venous blood samples will be collected by a qualified nurse from the antecubital vein into EDTA-treated vacutainers and centrifuged at 1500g for 10 minutes. Plasma will then undergo a second centrifugation at 2500g for 15 minutes and be stored in cryogenic vials at -80ºC. BDNF will be measured using the Human/Rat BDNF ELISA Kit (Proteintech Europe; sensitivity: 0.1 pg/mL; range: 12.5-800 pg/mL). PTau217 will be measured using the Human Phosphorylated Tau 217 ELISA Kit (GenoChem World; sensitivity: 0.1 pg/mL; range: 0.8-40 pg/mL).

SECONDARY OUTCOMES:
Physical activity levels | During one week prior to baseline
  An accelerometer (ActiGraph GT3X, Actigraph Corporation, Pensacola, FL) will be provided to all participants one week prior to the assessments to monitor physical activity levels during all waking hours, except during the shower or bath. Registration will take place over a seven-day period, including at least three weekdays (Monday through Friday) and two days during the weekend. The accelerometer will be positioned on the right hip of each participant through the use of an elastic belt. Their position will be reviewed before and after the registration period and participants will be provided with a diary to indicate the hours of use.
Sleep quality and cycle (objective) | During one week prior to baseline
  Participants will be provided with a Xiaomi® Smart Band 9 activity bracelet to monitor sleep quality. The device will record sleep cycle phases and data, as well as detailed data on heart rate and oxygen saturation.
Waist-hip ratio | Baseline
  Will be calculated using the waist circumference (in centimeters) and the hip circumference (in centimeters)
Hip circumference | Baseline
  Hip circumference will be assed in centimeters (cm)
Waist circumference | Baseline
  Waist circumference will be assed in centimeters (cm)
Sleep quality (subjective) | During one week prior to baseline
  Sleep quality will also be assessed by completing the Spanish version of the questionnaire Pittsburgh Sleep Quality Index (PSQI). This questionnaire consists of 24 items, of which 19 questions are self-assessed, while the remaining five are questions assessed by the patient's partner or roommate (the latter are not scored and are used only as clinical information). The total score ranges from 0-21 points, where a higher score indicates a worse subjective quality of sleep.
Heart rate variability | During one week prior to baseline
  By monitoring the heart rate of the participants, heart rate variability will be assessed, which involves the variation of the time intervals between beats (R-R intervals) and which is shown to be a useful tool in the control of the patient's health since it is an estimator of the balance between the activity of the sympathetic and parasympathetic autonomic nervous system . To evaluate heart rate variability, a polar H10 band and heart rate monitor (Polar Electro Oy, Kempele, Finland) and a mobile application, specifically Elite HRV will be used. Heart rate variability will be monitored daily for the week prior to the initial assessment visits. To do this, participants will be instructed to take the measurement the first 5 minutes as soon as they wake up and on an empty stomach.
Stress levels | Baseline
  The level of perceived stress will be assessed through the perceived stress questionnaire (PSQ). This questionnaire consists of 30 items and is carried out autonomously in the presence of the evaluator (score goes from 0 to 120 points, with higher score indicating more perceived stress levels). In addition, the Perceived Stress Scale (Perceived Stress Scale (PSS)) in its version of 14 items that are carried out in a self-administered way (score goes from 0 to 56, with higher scores indicating more stress levels).
Plasma testosterone/cortisol ratio | Baseline
  Plasma testosterone/cortisol ratio using ELISA kits. Fasting venous blood samples will be collected from the antecubital vein into EDTA-treated vacutainers and centrifuged at 1500g for 10 minutes. Plasma will then undergo a second centrifugation at 2500g for 15 minutes and be stored in cryogenic vials at -80ºC. Sample collection will be performed by a qualified nurse. Testosterone will be measured using the Invitrogen™ High Sensitivity Competitive ELISA Kit (Life Technologies; sensitivity: 2.97 pg/mL; range: 317.0-8440.5 pg/mL). Cortisol will be assessed with the Invitrogen™ Cortisol Competitive ELISA Kit (Life Technologies; sensitivity: 27.6 pg/mL; range: 8.5-23.8 µg/mL).
Nutritional habits | Baseline
  Adherence to the Mediterranean diet will be assessed through the Mediterranean Diet Quality Index in childhood and adolescence (KIDMED) questionnaire. This quiz It consists of 16 questions that evaluate adherence to this diet in children and young people (from 2 to 24 years old) and can be performed self-administered or conducted by an interviewer. The score goes from -4 to 12, with higher score indicating better adherence to Mediterranean diet.
Handgrip strength | Baseline
  Handgrip strength will be assessed using the hand-held Jamar® Plus Smart Dynamometer (Patterson Medical Ltd., Sammons Preston, Nottinghamshire, UK). Manual grip strength will be recorded on both limbs and the dynamometer will be adjusted to hand size prior to testing. The participant's elbow should be in 90° flexion and the forearm fully supported on a table.
Gas exchange analysis | Baseline
  The values of mean and peak gas exchange (ml·kg-1·min-1) during a stress test. The gas analyzer that will be used in this study (Cortex Metalyzer 3B, Leipzig, Germany).
  The basal metabolic rate (ml·kg-1·min-1) will be determined by recording the variables mentioned above for 15 minutes in supine position.
Cardiovascular response | Baseline
  The values of mean and peak heart rate (beats per minute) will be assessed using a polar H10.
Excess Post-exercise Oxygen Consumption | Baseline
  The Excess Post-exercise Oxygen Consumption (EPOC) post-exercise will be recorded on ml·kg-1·min-1. This will be calculated every minute for 12 min after the end of the exercise.
Weight | Baseline
  Weight will be assess on kilograms (kg)
Height | Baseline
  Height will be assess on centimeters (cm)
Body surface area | Baseline
  Weight and height will be combined to report body surface area (BSA) in kg·cm-1
Bioimpedance | Baseline
  The NUTRILAB bioimpedance device (AKERN Srl, Florence, Italy) will be used. This non-invasive method measures the body's resistance and reactance of the body to the passage of a low-intensity electric current and enables the determination of various body parameters. Bioimpedance provides accurate data on body composition. Users will be instructed to remove all metal-containing objects and remain in a supine position on a couch during the measurements, with the legs in 45° abduction, the shoulders in 30° abduction relative to the center of the body and the hands in pronation. After cleaning the skin with alcohol, two adhesive electrodes (Biatrodes Akern Srl, Florence, Italy) will be placed on the surface of the right hand and two on the right foot. The measurement results will be given in different unit measures depending on the specific variable assessed.
Cognitive performance | Baseline
  Cognitive performance will be assessed through the questionnaire Frontal Assessment Battery (FAB). This questionnaire allows for rapid assessment of executive function through six tests that correspond to each specific cognitive or behavioral domain related to the frontal lobes. The scores ranges from 0 to 18 where higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lista, PhD, Principal Investigator — Miguel de Cervantes European University; Susana López-Ortiz, PhD, Study Chair — Miguel de Cervantes European University
Locations (1):
- Miguel de Cervantes European University, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurtado-Pomares M, Juarez-Leal I, Company-Devesa V, Sanchez-Perez A, Peral-Gomez P, Espinosa-Sempere C, Valera-Gran D, Navarrete-Munoz EM. Psychometric properties of the Spanish version of the Frontal Assessment Battery (FAB-E) and normative values in a representative adult population sample. Neurologia (Engl Ed). 2024 Oct;39(8):694-700. doi: 10.1016/j.nrleng.2022.09.004. Epub 2022 Oct 7. PMID 36216225
- [Background] Benito PJ, Alvarez-Sanchez M, Diaz V, Morencos E, Peinado AB, Cupeiro R, Maffulli N; PRONAF Study Group. Cardiovascular Fitness and Energy Expenditure Response during a Combined Aerobic and Circuit Weight Training Protocol. PLoS One. 2016 Nov 10;11(11):e0164349. doi: 10.1371/journal.pone.0164349. eCollection 2016. PMID 27832062
- [Background] Jarvinen L, Lundin Petersdotter S, Chaillou T. High-intensity resistance exercise is not as effective as traditional high-intensity interval exercise for increasing the cardiorespiratory response and energy expenditure in recreationally active subjects. Eur J Appl Physiol. 2022 Feb;122(2):459-474. doi: 10.1007/s00421-021-04849-4. Epub 2021 Nov 19. PMID 34799752
- [Background] Perrotta AS, Jeklin AT, Hives BA, Meanwell LE, Warburton DER. Validity of the Elite HRV Smartphone Application for Examining Heart Rate Variability in a Field-Based Setting. J Strength Cond Res. 2017 Aug;31(8):2296-2302. doi: 10.1519/JSC.0000000000001841. PMID 28195974
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Concheiro-Moscoso P, Groba B, Alvarez-Estevez D, Miranda-Duro MDC, Pousada T, Nieto-Riveiro L, Mejuto-Muino FJ, Pereira J. Quality of Sleep Data Validation From the Xiaomi Mi Band 5 Against Polysomnography: Comparison Study. J Med Internet Res. 2023 May 19;25:e42073. doi: 10.2196/42073. PMID 37204853
- [Background] Klein AB, Williamson R, Santini MA, Clemmensen C, Ettrup A, Rios M, Knudsen GM, Aznar S. Blood BDNF concentrations reflect brain-tissue BDNF levels across species. Int J Neuropsychopharmacol. 2011 Apr;14(3):347-53. doi: 10.1017/S1461145710000738. Epub 2010 Jul 7. PMID 20604989
- [Background] Poo MM. Neurotrophins as synaptic modulators. Nat Rev Neurosci. 2001 Jan;2(1):24-32. doi: 10.1038/35049004. PMID 11253356
- [Background] Gomez-Pinilla F, Tyagi E. Diet and cognition: interplay between cell metabolism and neuronal plasticity. Curr Opin Clin Nutr Metab Care. 2013 Nov;16(6):726-33. doi: 10.1097/MCO.0b013e328365aae3. PMID 24071781
- [Background] Walsh R. Lifestyle and mental health. Am Psychol. 2011 Oct;66(7):579-92. doi: 10.1037/a0021769. PMID 21244124